CLINICAL TRIAL: NCT04972903
Title: Impact of Malnutrition on Pharmacokinetic of Rifampicin, Isoniazid, Pyrazinamide and Ethambutol in TB-HIV Co-infected Children
Brief Title: Impact of Malnutrition on Pharmacokinetic of Rifampicin, Isoniazid, Pyrazinamide and Ethambutol in TB-HIV Co-infected Children (TB-Speed TB-PK)
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Agency for Research on AIDS and Viral Hepatitis (ANRS) (Other)
Responsible Party: Sponsor
Other Study IDs: C20-17
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis; Pulmonary
Keywords: HIV; Childhood tuberculosis; Severe acute malnutrition; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Tuberculosis; Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1.HIV+/SAM+: Group 1. HIV-infected with SAM (WHZ<-3SD or edematous malnutrition or MUAC <115) (HIV+/SAM+)
- Group 2. HIV+/SAM-: Group 2. HIV-infected without SAM (none of the 3 criteria above) (HIV+/SAM-)
- Group 3. HIV-/SAM+: Group 3. HIV-negative with SAM (WHZ<-3SD or edematous malnutrition or MUAC <115) (HIV-/SAM+)
- Group 4. HIV-/SAM-: Group 4. HIV-negative without SAM (none of the 3 criteria above) (HIV-/SAM-)

SUMMARY:
TB-Speed TB-PK is a cross-sectional PK study of anti-TB treatment nested in the TB-Speed HIV and TB-Speed SAM studies aiming at assessing the impact of malnutrition on PK of rifampicin, isoniazid, pyrazinamide, and ethambutol in TB-HIV co-infected children in Uganda and Zambia.

DETAILED DESCRIPTION:
Tuberculosis can worsen malnutrition and in turn malnutrition increases the risk of TB. HIV infection is prevalent in children with TB and SAM and is often associated with poor outcomes when present. TB alone is the leading cause of death of among HIV-infected children worldwide accounting for a third of all the death in this group.

In 2010, the WHO recommended increased dose for rifampicin (+50%), isoniazid (+100%), and pyrazinamide (+33%) based on PK data showing that plasma drug concentrations in children using standard adult dosages did not reach target levels. In children that are TB/HIV co-infected, drug-drug interactions between anti-TB drugs and antiretroviral drugs are of concern.

The investigators hypothesize that HIV-infection and SAM, each one on its own, may have an impact on TB drugs concentrations. Furthermore, SAM is frequent in children with HIV, and may affect the metabolism of anti-TB drugs and consequently result in low serum concentration.

TB-Speed TB-PK is a cross-sectional PK study of anti-TB treatment nested in the TB-Speed HIV and TB-Speed SAM studies aiming at assessing the impact of malnutrition on PK of rifampicin, isoniazid, pyrazinamide, and ethambutol in TB-HIV co-infected children. It will be implemented in Uganda and Zambia. Children will also be enrolled from routine care for TB outside of the TB- Speed HIV and TB-Speed SAM studies.

ELIGIBILITY:
INCLUSION CRITERIA:

* Gr1. HIV-infected children with SAM

  * Age 6 months to 5 years
  * Diagnosed with TB and first line TB treatment to be initiated or started less than 4 weeks prior to inclusion
  * HIV-infection
  * SAM as defined by WHO at the time of starting TB treatment
  * Weight-for-height z-score (WHZ) < -3 SD,
  * OR MUAC <11.5 cm or
  * OR presence of bilateral pitting oedema of nutritional origin
  * Ability to take drugs orally during the planned PK day
  * Signed informed consent from parents or guardian
* Gr2. HIV-infected children without SAM

  * Age 6 months to 5 years
  * Diagnosed with TB and first line TB treatment to be initiated or started less than 4 weeks prior to inclusion
  * HIV-infection
  * Absence of SAM as defined by WHO at the time of starting TB treatment
  * Weight-for-height z-score (WHZ) > -3 SD,
  * AND MUAC >11.5 cm or
  * AND absence of bilateral pitting oedema of nutritional origin
  * Ability to take drugs orally during the planned PK day
  * Signed informed consent from parents or guardian
* Gr3. HIV-negative children with SAM

  * Age 6 months to 5 years
  * Diagnosed with TB and first line TB treatment to be initiated or started less than 4 weeks prior to inclusion
  * HIV-negative
  * SAM as defined by WHO at the time of starting TB treatment
  * Weight-for-height z-score (WHZ) < -3 SD,
  * OR MUAC <11.5 cm or
  * OR presence of bilateral pitting oedema of nutritional origin
  * Ability to take drugs orally during the planned PK day
  * Signed informed consent from parents or guardian
* Gr4. HIV-negative children without SAM

  * Age 6 months to 5 years
  * Diagnosed with TB and first line TB treatment to be initiated or started less than 4 weeks prior to inclusion
  * HIV-negative
  * Absence of SAM as defined by WHO at the time of starting TB treatment
  * Weight-for-height z-score (WHZ) > -3 SD,
  * AND MUAC >11.5 cm or
  * AND absence of bilateral pitting oedema of nutritional origin
  * Ability to take drugs orally during the planned PK day
  * Signed informed consent from parents or guardian

NON INCLUSION CRITERIA:

* Very ill or moribund children unable to take drugs orally or requiring nasogastric drug intake
* Severe anaemia (Hb < 6 g/dl),
* Severe renal impairment (DAIDS grade 3 and above)
* Severe hepatic impairment (DAIDS grade 3 and above)
* Children on second line TB drugs

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Intensive PK of rifampicin, isoniazid, pyrazinamide, and ethambutol will be performed between 2 to 4 weeks of TB treatment in the following 4 groups of children receiving first-line anti-TB treatment:
  * Group (Gr) 1. HIV-infected with SAM (WHZ<-3SD or edematous malnutrition or MUAC <115) (HIV+/SAM+)
  * Gr2. HIV-infected without SAM (none of the 3 criteria above) (HIV+/SAM-)
  * Gr3. HIV-negative with SAM (WHZ<-3SD or edematous malnutrition or MUAC <115) (HIV-/SAM+)
  * Gr4. HIV-negative without SAM (none of the 3 criteria above) (HIV-/SAM-)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Effect of SAM on Peak plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB | 6 months
  Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol peak concentration (Cmax)
Effect of SAM on minimum plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB | 6 months
  Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol minimum concentration (Cmin or C trough)
Effect of SAM on Area Under the Curve plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB | 6 months
  Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol exposure (Area Under the Curve - AUC)

SECONDARY OUTCOMES:
Effect of HIV-infection and antiretroviral treatment on Peak plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB and SAM | 6 months
  Cmax of Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol in children with HIV infection on or off ART and children without HIV infection
Effect of HIV-infection and antiretroviral treatment on Minimum plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB and SAM | 6 months
  Cmin of Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol in children with HIV infection on or off ART and children without HIV infection
Effect of HIV-infection and antiretroviral treatment on Area Under the Curve plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol in children with TB and SAM | 6 months
  AUC of Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol in children with HIV infection on or off ART and children without HIV infection
WHO-based dosages will achieve rifampicin, isoniazid, pyrazinamide, and ethambutol drug concentrations above the target therapeutic concentrations in HIV-TB co-infected children with and without SAM | 6 months
  Proportion of children with AUC24 and Cmax above the recommended threshold for Rifampicin, Isoniazid, Pyrazinamide, and Ethambutol
Effect of personnal parameters (nutritional parameters, HIV-infection, antiretroviral treatment, age, liver enzymes and NAT2 status) on CL/F of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB | 6 months
  CL/F(Apparent total clearance of the drug from plasma) after oral administration of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB.
Effect of personnal parameters (nutritional parameters, HIV-infection, antiretroviral treatment, age, liver enzymes and NAT2 status) on V/F of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB | 6 months
  V/F (Apparent volume of distribution after administration) after oral administration of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB.
Effect of personnal parameters (nutritional parameters, HIV-infection, antiretroviral treatment, age, liver enzymes and NAT2 status) on Ka of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB | 6 months
  Ka (Absorption rate constant) after oral administration of rifampicin, isoniazid, pyrazinamide, and ethambutol in HIV-infected children with TB.
Relationship between all-cause mortality in children with TB and SAM, and Peak plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol. | 6 months
  Define the best Cmax plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol for treatment sucess.
Relationship between all-cause mortality in children with TB and SAM, and the minimum plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol. | 6 months
  Define the best Cmin plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol for treatment sucess.
Relationship between all-cause mortality in children with TB and SAM, and Area Under the Curve plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol. | 6 months
  Define the best AUC plasma concentration of rifampicin, isoniazid, pyrazinamide, and ethambutol for treatment sucess.
Rifampicin protein binding in relation with malnutrition and albuminemia | 6 months
  Proportion of protein bound rifampicin in children with SAM and association with albuminemia

CONTACTS AND LOCATIONS:
Locations (4):
- Uganda (2):
  - Mulago National Referral Hospital, Kampala
  - Mbarara Regional Hospital, Mbarara
- Zambia (2):
  - The University Teaching Hospital, Lusaka
  - Arthur Davison Children Hospital, Ndola

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TB-Speed project official website — http://www.tb-speed.com